CLINICAL TRIAL: NCT05337826
Title: Readiness, Education, and Sustainability for CGM Technology Adoption Model for Older Adults With Insulin-treated Diabetes
Brief Title: The REST Study for CGM Use in Older Adults With Insulin-treated Diabetes
Acronym: REST
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: State University of New York - Upstate Medical University (Other); Cecilia Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000174
Record Dates: First submitted 2022-04-05; First posted 2022-04-20 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus
Keywords: older adults; CGM; diabetes technology; telehealth
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental)
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Participants will enroll in a series of remote educational visits conducted by CDCES to assess readiness and barriers to CGM initiation and utilization, with the goal to sustain use of CGM Technology over time in older populations on complex insulin regimen.
  Other Names: the REST model

SUMMARY:
To assess the efficacy of the REST model in facilitating adoption and sustained use of CGM, in older adults with Type 1 diabetes (T1D) or Type 2 Diabetes (T2D) on complex insulin regimens. To examine barriers and enablers for the implementation feasibility of the REST intervention model using a mixed-methods approach. To assess the impact of REST model on economic factors and quality of life measures. The goal of this study is to facilitate the adoption of continuous glucose monitoring (CGM) in older adults (≥65 years) with diabetes mellitus (DM) on complex insulin regimens, and additionally, to build a framework for sustained CGM use over time using a novel patient-centered model - the REST model.

DETAILED DESCRIPTION:
Older adults with diabetes on multiple insulin injections are at greater risk of hypoglycemia and its poor outcomes. Use of continuous glucose monitoring (CGM) has shown to improve glycemic control and reduce hypoglycemia in this age group. Despite Medicare coverage for CGM, uptake in this age group is still low. The goal of this study is to facilitate the adoption of continuous glucose monitoring (CGM) in older adults (≥65 years) with diabetes mellitus (DM) on complex insulin regimens, and additionally, to build a framework for sustained CGM use over time using a novel patient-centered model - the REST model. This model will assess Readiness and barriers to CGM initiation and utilization, provide remote Education, and implement a framework for Sustainability of CGM Technology adoption. The study will assess the impact of the REST model and its ability to increase CGM uptake and use in this age group, as well as its effectiveness on improving glycemic metrics. The study will also evaluate the impact of the REST model on economic and health-related quality-of-life measures.

ELIGIBILITY:
Inclusion Criteria:

* Older adults age ≥65 years
* T1D or T2D with duration longer than 1 year
* Insulin treatment includes: ≥3 insulin injections/day or on insulin pump therapy
* CGM naïve and/or CGM users (Dexcom G6) who are not meeting glycemic goals (per

CGM metrics):

* ≥4% hypoglycemia (sensor glucose ≤70 mg/dL) or
* time in range (70-180 mg/dL) TIR ≤40 %
* Willing to wear CGM Dexcom at all times while in the study
* Willing to use/carry personal or loaned smart phone device to use as Dexcom receiver for continual data upload to cloud

Exclusion Criteria:

* Life expectancy <1 year
* End-stage renal disease (eGFR< 30ml/min)
* On acetaminophen >4 gr/day due to interference with Dexcom G6 sensor readings
* On hydroxyurea therapy due to interference with Dexcom G6 sensor readings
* Impaired vision and hearing which would interfere with participation in remote video visits
* Use of hybrid closed-loop systems (this may require different and additional focused education and will not be addressed in this study).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
The co-primary effectiveness outcomes | Baseline to 6 months
  Change in time spent in hypoglycemia (sensor glucose <70 mg/dL and ii) Change in individualized Time in Range goal
The co-primary implementation outcomes | Baseline vs 6 months
  Change in adoption of CGM by remote education (change in number of CGM users and ii) change in number of hours of CGM use per week

SECONDARY OUTCOMES:
Visits to maintain CGM use | 6 months
  Total time spent and the number of remote and in-person visits needed to initiate and maintain CGM use
Visits to maintain CGM use | Month 12
  Total time spent and the number of remote and in-person visits needed to initiate and maintain CGM use
Resource utilization | Baseline vs 6 months
  Change in resource utilization (episodes of severe hypoglycemia, emergency department visits, and hospitalizations)
Resource utilization | 6 months vs 12 months
  Change in resource utilization (episodes of severe hypoglycemia, emergency department visits, and hospitalizations)
Time spent in hypoglycemia | 6 months vs 12 months
  Change in time spent in hypoglycemia ( sensor glucose <70 mg/dL)
Cost effectivness | 6 months
  Cost-effectiveness ratios to assess the economic aspects for REST model compared standard of care
Cost Effectivness | 12 months
  Cost-effectiveness ratios to assess the economic aspects for REST model compared standard of care
Diabetes health related quality of life measures | Baseline vs 6 months
  Change in quality of life measures (diabetes distress, hypoglycemia fear, EQ-5D)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Joslin Diabetes Center, Boston, Massachusetts
  - SUNY Upstate Medical University, Syracuse, New York

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices) will be shared to Researchers who provide a methodologically sound proposal, to achieve the aims in the approved proposal.
Supporting Information: Study Protocol
Time Frame: Start 6 months after publication and end 5 years after publication
Access Criteria: Proposals should be directed to elena.toschi@joslin.harvard.edu. To gain access, data requestors will need to sign a data access agreement.